CLINICAL TRIAL: NCT04071470
Title: Increasing Family-based Support for PrEP Adherence Among Discordant Couples Through Storytelling
Brief Title: Storytelling to Increase Family Support for Pre Exposure Prophylaxis Use
Acronym: PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Friends in Global Health (Other)
Responsible Party: Principal Investigator, Carolyn Audet, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: storytelling
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: We will be comparing standard of care PrEP services with a storytelling intervention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care for pregnant women at risk of HIV seroconversion includes couples counseling and access to PrEP (women) and ART (men)
  Interventions: Drug: PrEP
- Storytelling Intervention (Experimental): Participants in this group will receive the same services as those in the SOC but will also be provided three storytelling sessions for themselves and their families as a way to educate and de-stigmatize PrEP services.
  Interventions: Behavioral: Storytelling; Drug: PrEP

INTERVENTIONS:
Behavioral: Storytelling — Couples in the storytelling intervention will receive 3 storytelling sessions- the couple can include any family or friends who they feel could support them during their treatment. Stories will include stories of couples who are supportive, those who experience difficulties, and families who do/do not support their use of PrEP
  Arms: Storytelling Intervention
Drug: PrEP — Patients at risk of HIV acquisition will be provided PrEP medications and counseling in ANC

SUMMARY:
Pre-exposure prophylaxis (PrEP) is highly effective at preventing HIV infection but requires high levels of medication adherence, particularly among women. The purpose of this proposal is to evaluate the clinical impact and mechanisms of a family-based storytelling intervention (vs. couples counseling) to improve PrEP adherence and retention among at-risk pregnant/lactating women and their HIV-infected male partners in rural Mozambique. This potentially high impact intervention provides the opportunity to test a culturally relevant approach to PrEP engagement; if proven feasible and effective, family-based storytelling for PrEP engagement could be adopted to reduce HIV incidence among pregnant/lactating women and eliminate mother-to-child transmission (MTCT).

DETAILED DESCRIPTION:
Project Summary: Pregnancy and the postpartum period are associated with an increased risk of HIV acquisition. HIV acquisition is of particular concern during pregnancy and while the mother is breastfeeding given the associated increased risk of mother-to-child transmission (MTCT). Approximately 10% of pregnant women attending antenatal care (ANC) in Mozambique are in serodiscordant relationships (HIV-negative woman/ HIV-positive man). High rates of MTCT (14%; 12,000 infants/ year) may be affected by the high rate at which pregnant women seroconvert after their first ANC visit. Beginning in 2018, pre-exposure prophylaxis (PrEP) was available to serodiscordant couples, yet only 44% of pregnant women were retained in care at 3 months.

Our current R01-funded project, Partners-based HIV Treatment for Seroconcordant Couples (R01MH113478), is testing a couple-based intervention for HIV-positive expectant parents living in extremely rural communities. Our Men for Health intervention ("Homens para Saúde+"- HoPS+) consists of (1) couple-based HIV care and treatment; (2) couple-centered education; and (3) expert-patient support. Preliminary data the HoPS+ study suggest that couple-based counseling and education is more successful at reducing maternal depression than individual care. However, couple-based sessions have not led to significantly greater improvements in HIV knowledge or social support. Given the importance of these factors on treatment adherence, this grant would allow us to revise the peer engagement strategy to increase knowledge transfer and engender partner support.

The investigators propose testing the impact of a peer-delivered oral storytelling intervention to increase retention in, and adherence to, PrEP/ART among expectant serodiscordant couples. People are 7 times more likely to remember a story compared to facts alone. Couples are also highly influenced by their immediate and extended families; >95% of patients disclose their HIV status to members of their family. The investigators hypothesize that the use of oral storytelling will facilitate learning and encourage family support and advocacy. The investigator will compare this model to couple-based education and counseling. This innovative intervention tests a culturally relevant approach to improve ART/PrEP delivery. The investigators propose a rigorous individually randomized controlled trial at one of our current HoPS+ sites where 11% of expectant couples were serodiscordant in 2018. The investigators will randomize 70 HIV-uninfected pregnant women and 70 of their HIV-infected partners (total 140) to either the intervention or control condition.

The Specific Aims of this study are: (1) Compare the effect of a storytelling intervention (vs. couples-based counseling) on participant knowledge, motivation, and behavioral skills associated with PrEP retention and adherence; and (2) Evaluate the impact of a storytelling intervention on adherence to PrEP/ART medications. Our team of Mozambican and U.S. investigators has a proven record of international HIV research success, specific recent experience with partner-based HIV and PrEP delivery, and experience with the use of theater/storytelling to change HIV-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women/male partner

1. Discordant couple, one pregnant woman (HIV-) and her HIV+ male partner
2. Both persons must agree to take PrEP (pregnant woman)/ART (male partner)
3. The woman's due date is >4 weeks from study enrollment
4. Both persons must be 18 years or older
5. Both persons (parents) must be willing to consent to an infant record search
6. Neither member of the couple can be under the influence of alcohol at the time of consent.

Family members of expectant couple

1. Must be a relative living in the participants household or living in the study community
2. Must agree to participate in at least one of the storytelling sessions;
3. Must be 18 years of age or older
4. Must not be under the influence of alcohol
5. Must be willing to participate in the interview.

Exclusion Criteria:

Pregnant woman/Male Partner

1. One member of the couple is unwilling to enroll in treatment

Family members

1. Unable to attend storytelling session
2. Expectant couple expresses unwillingness for the family member to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Minisitry of Health Health Facility, Quelimane, Zambezia Province, Mozambique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sack DE, De Schacht C, Paulo P, Graves E, Emilio AM, Matino A, Fonseca CL, Aboobacar AU, Van Rompaey S, Audet CM. Pre-exposure prophylaxis use among HIV serodiscordant couples: a qualitative study in Mozambique. Glob Health Action. 2021 Jan 1;14(1):1940764. doi: 10.1080/16549716.2021.1940764. PMID 34229580

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Storytelling Intervention
Started | 62 | 66
Completed | 62 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Storytelling Intervention | Total
Number analyzed (Participants) | 62 | 66 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (5.59) | 25.8 (6.64) | 25.1 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 31 | 33 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 66 | 128
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Occupation [Count of Participants; unit: Participants]
  Merchant | 10 | 6 | 16
  Domestic | 23 | 26 | 49
  Farmer | 22 | 21 | 43
  Fisherman | 0 | 1 | 1
  Other | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Adherence to PrEP Medication
Description: Maternal adherence to medication as measured via monthly medication pick up records
Time Frame: 3 months
Population: We only looked at PrEP use among the women in the study
Measure: Median (Inter-Quartile Range); unit: percentage of pills taken daily
Arm/Group | Standard of Care | Storytelling Intervention
Number analyzed (Participants) | 31 | 33
percentage of pills taken daily | 96.6 [80.6 to 100] | 95.5 [78.1 to 98.9]

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Intervention Arm: Received the three storytelling sessions
- Control Arm: Received only standard of care services
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/62
Other Adverse Events (participants affected / at risk) | 0/66 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT04071470/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT04071470/ICF_001.pdf